CLINICAL TRIAL: NCT01982461
Title: A Randomized, Open-label, Active-controlled Study to Evaluate the Efficacy and Safety of Roty F.C. Tablets 10mg Versus Crestor 10mg F.C. Tablets in Patients With Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy and Safety of Rosuvastatin in Hypercholesterolemia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pin Siang Medical Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSMB102ROS10-01
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): One Rosuvastatin tablet 10mg taken once daily.
  Interventions: Drug: Rosuvastatin
- Crestor® (Active Comparator): One Crestor® tablet 10mg taken once daily.
  Interventions: Drug: Crestor®

INTERVENTIONS:
Drug: Rosuvastatin — 10mg,once daily
  Other Names: Roty
  Arms: Rosuvastatin
Drug: Crestor® — 10mg,once daily
  Other Names: Rosuvastatin
  Arms: Crestor®

SUMMARY:
The objective of this trial is to assess the efficacy of reducing plasma low-density lipoprotein(LDL) cholesterol and safety in two different brand drugs, Roty F.C. Tablets 10mg and Crestor 10mg F.C. Tablets in hypercholesterolemia population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20 to 85;
* LDL - C between 130 mg/dL and 250 mg/dL;
* TG < 400 mg/dL;
* Who without use of any statin within 2 week prior to the trial;
* Informed consent given.

Exclusion Criteria:

* Known hypersensitivity or history of SAE with another HMG-CoA reductase inhibitor, in particular any history of myopathy;
* Active liver disease/severe hepatic impairment(Child-Pugh C,ALT2×ULN);
* Treatment with Cyclosporin or any disallowed drug;
* Patients with unstable angina pectoris;
* Pregnant, lactating women;
* Patients who have severe medical condition(s) that in the view of the Investigator prohibits participation in the trial.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable will be defined as the percent mean change in LDL-C from baseline to 12 weeks. | baseline to week 12

SECONDARY OUTCOMES:
The secondary efficacy variable will be described as the change of plasma AGE, sRAGE, Gas6 and sAx1. | baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Hung, M.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan